CLINICAL TRIAL: NCT02359500
Title: Safety and Efficacy Study of 68Ga-Dotatoc Positron Emission Tomography for Diagnosis for Staging, Restaging and Assessment of Response to Treatment in Somatostatin Receptor-Positive Neuroendocrine Tumors
Brief Title: 68Ga-Dotatoc Positron Emission Tomography (PET) for Somatostatin Receptor-Positive Neuroendocrine Tumors (NETs)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: compound no longer available
Sponsor: Lale Kostakoglu (Other)
Responsible Party: Sponsor-Investigator, Lale Kostakoglu, Chief of Nuclear Medicine and Molecular Imaging, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GCO 14-2008
Record Dates: First submitted 2015-01-23; First posted 2015-02-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Neuroendocrine Tumors; Carcinoid Tumors
Keywords: 68Ga- DOTATOC; Diagnosis; Somatostatin Receptor-Positive Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoid Tumor; Disease | interventions — Ga(III)-DOTATOC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTATOC PET (Experimental): patients with known or suspected somatostatin receptor positive neuroendocrine tumors (NETs)
  Interventions: Drug: 68Ga-DOTATOC PET

INTERVENTIONS:
Drug: 68Ga-DOTATOC PET — 68Ga-DOTATOC as a diagnostic PET/CT imaging agent for the detection of NETs, mainly carcinoid tumors.
  Other Names: [68Ga]-DOTA-tyr3-Octreotide; [68Ga]-DOTATOC

SUMMARY:
This study plans to demonstrate the safety and efficacy of [68Ga]-DOTA-tyr3-Octreotide ([68Ga]-DOTATOC) as an accurate imaging technique for diagnosis, staging, and monitoring of response to treatment in patients with Somatostatin receptor expressing tumors who undergo imaging with a clinical indication. The investigators will conduct a study for 68Ga-DOTATOC as a diagnostic PET/CT imaging agent for the detection of NETs, mainly carcinoid tumors. 68Ga-DOTATOC will be used in diagnostic assessment of patients with known or suspected NETs for whom there is an appropriate standard clinical indication for 68Ga-DOTATOC PET/CT either at staging or during follow up.

DETAILED DESCRIPTION:
Rationale and overall study design This study is planned to demonstrate the safety and efficacy of [68Ga]-DOTA-tyr3-Octreotide ([68Ga]-DOTATOC) as an accurate imaging technique for diagnosis, staging, and monitoring of response to treatment in patients with Somatostatin receptor expressing tumors who undergo imaging with a clinical indication.

Neuroendocrine tumors (NET) are rare neoplasms of neuroendocrine origin. Neuroendocrine tumors are solid malignant tumors that arise from dispersed neuroendocrine cells found throughout the body. They are well known for their heterogeneity which makes it difficult to obtain uniform clinical data and establish universal guidelines for the diagnosis and treatment of NETs. NETs are characterized by overexpression of somatostatin receptors, which can be visualized and targeted by radiolabeled somatostatin analogues. 111In-diethylenetriaminepentaacetic acid-octreotide scintigraphy (111In-Octreotide) with single photon emission tomography (SPECT) is currently the standard imaging modality for evaluating patients with NETs. 111In Octreotide is the only FDA approved radiopharmaceutical available on the market for assessing the extent of involvement by NETs at both staging and follow up periods. However, the sensitivity of this imaging modality is lower compared to the positron emission tomography (PET) radiotracer 68Ga-DOTA0-Tyr3]octreotide (68Ga-DOTA-TOC). Based on the improved sensitivity, 68Ga DOTATOC PET leads to significant changes in 30% of patients. Importantly, the radiation exposure of 68Ga-DOTATOC PET is lower than that of 111In Octreotide and also the imaging with 68Ga-DOTATOC PET scan yields fast read-outs on the same day compared to 24-48 hour read-outs with 111In Octreotide scan. These advantages make the 68Ga labeled somatostatin analog more attractive from both the patient and management perspectives. The improved resolution and quantitation of uptake obtained with Ga-68 DOTATOC PET should provide a more accurate assessment of somatostatin receptor density, which will lead to a more accurate prediction of treatment response to somatostatin analogues.

While the investment costs for the scanner, the radiochemistry equipment are higher for 68Ga-DOTATOC PET/CT compared with 111In-DTPA-octreotide scintigraphy and SPECT, with the provision of this imaging molecule by an established commercial radiopharmaceutical company that in with compliance to FDA 21 CFR Part 212 IBA Molecular Inc, NJ, USA, this will not pose a limitation for the Mount Sinai Medical Center. In this setting, 68Ga-DOTATOC PET/CT production and personnel costs will be borne by the commercial entity, however, Mount Sinai Medical Center will purchase the 68Ga-DOTATOC based on a per patient schedule. Since this imaging modality does not have a quote for reimbursement by the insurance carriers, the imaging cost is considered a potential burden on the patient until it is approved by the U.S. Food and Drug Administration (FDA). There is significant amount of European based clinical data (>1000 patients) to prove the safety and efficacy of this imaging agent, therefore, a phase II or III clinical trial in the US is redundant and will only delay the approval of this imaging probe. Recently, Ga-68 DOTATOC has been designated as an orphan drug by the FDA for the management of NET. This designation will probably lead to faster approval of the agent, which would greatly benefit NET patients in the US. Currently, there are only several small U.S.-based clinical trials for Ga-68 labeled NET PET agents available for patients; otherwise they must travel out of the country if the scan is required to manage their disease.

The investigators, therefore, aim to provide this superior imaging technique to NET patients for better disease management by the referring physicians, however, this objective cannot be attained unless at least a partial funding mechanism exists to make it affordable by the patients until the approval of this superior imaging probe. In this regard, the investigators are aiming at recovering the cost of the radiotracer from the local insurance carrier through the cost recovery system.

Participant Enrollment Participants will be recruited from the Mount Sinai Medical Center. Participants who will be approached regarding the study are those individuals who are being seen for known or suspected malignancies.

Patients may remain on their somatostatin therapies throughout the study with no management change merely based on the 68Ga -DOTATOC PET/CT imaging findings. The management of these patients will be based on the standard of care and any change will be at the discretion of the referring physician. All pertinent dosing information must be collected and reported.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected somatostatin receptor positive NETs (e.g. carcinoid, pancreatic neuroendocrine tumors, and pheochromocytoma). Supporting evidence may include MRI, CT, biochemical markers, and or pathology report.
* Karnofsky performance status of ≥50 (or ECOG/WHO equivalent)
* Off Sandostatin (octreotide acetate)-long acting release (LAR) > 4 weeks and off immediate release (subcutaneous) for at least 12 hrs prior to 68Ga-DOTATOC PET-CT imaging
* Able to provide informed consent
* At least 18 years of age

Exclusion Criteria:

* Pregnancy or breast feeding. A negative serum pregnancy test is required for all female subjects with child- bearing potential
* Surgical resection, chemotherapy, radiation therapy, or biologic therapy since last Octreoscan + CT; continuation of the same dose of Sandostatin-LAR or subcutaneous Sandostatin is allowed
* Medical condition uncontrolled by treatment making completion of study unlikely
* Patients exceeding the weight limitations of the scanner or are not able to enter the bore of the PET/CT scanner due to Body Mass Index (BMI)
* Inability to complete the needed investigational and standard-of-care imaging examinations due to other reasons (e.g. severe claustrophobia)
* Any additional medical condition, serious intercurrent illness or other extenuating circumstance that, in the opinion of the Investigator, may significantly interfere with study performance or interpretation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Change in size of lesion | baseline and 1 month
  Change in size of lesion at 1 month as compared to baseline

SECONDARY OUTCOMES:
Incidence of new lesions | baseline and 1 month
  Number of new lesions at 1 month as compared to baseline
Incidence of change in treatment | baseline and 1 month
  Change in treatment caused by result of 68Ga-DOTATOC PET/CT at 1 month as compared to baseline
Incidence of previously unknown primary tumor | baseline and 1 month
  Incidence of identification of the location of a previously unknown primary tumor at 1 month as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Lale Kostakoglu, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States